CLINICAL TRIAL: NCT03670667
Title: The Risk of Cancer Associated With the Use of Abatacept and Other Biologic Agents Among Rheumatoid Arthritis Patients
Brief Title: A Study to Determine the Risk of Cancer in Rheumatoid Arthritis (RA) Patients Who Use Abatacept and Other Biologic Agents
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM101-674
Record Dates: First submitted 2018-09-07; First posted 2018-09-13 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- RA patients treated with abatacept
  Interventions: Other: Non-Interventional
- RA patients treated with anti-TNFi's
  Interventions: Other: Non-Interventional
- RA patients treated with other biologics
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — Non-Interventional
  Groups: RA patients treated with abatacept
Other: Non-Interventional — Non-Interventional
  Groups: RA patients treated with anti-TNFi's
Other: Non-Interventional — Non-Interventional
  Groups: RA patients treated with other biologics

SUMMARY:
An observational study to determine the risk of cancer associated with the use of abatacept and other biologic agents among rheumatoid arthritis patients

ELIGIBILITY:
Inclusion Criteria:

* RA patients will be identified using algorithms that require ≥ 1 rheumatologist (physician specialty code: 66) diagnosis codes for RA (at least one of the following ICD9 diagnosis codes: 714.0, 714.2, 714.81) at any time before the first claim for a specific drug (Index date) during the study period and ≥1 physician (affiliated with physician evaluation & management codes, listed in the appendix 2) diagnosis codes within 12 months before the first claim for a specific drug use. The index date is defined as the date of the first claim for a specific drug use, and the baseline period is defined as 12 months prior to specific drug use
* Naive users of biologics, including abatacept, anti-TNFs (i.e. etanercept, adalimumab, certolizumab, golimumab, infliximab), rituximab, and tocilizumab, will be defined specific to each drug as no claim for that therapy in any time prior to the index date
* Eligible subjects, including cancer patients in SEER and non-cancer beneficiaries from 5% sample, must have been continuously enrolled in Medicare Parts A, B and D and not C at their index date and during baseline

Exclusion Criteria:

* Patients diagnosed with any cancer (ignoring non-melanoma skin cancer, which is not captured within SEER) before the use of biologics under study. Cancer cases will be identified based on the records in SEER
* Patients who were younger than 18 years on the index date
* Patients with claims for other types of auto-immune diseases (e.g. psoriatic arthritis, systemic lupus erythematosus) during baseline
* Month or year of diagnosis of malignancy in SEER was unknown
* Cancer cases who were identified by death certificate or autopsy only in SEER

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will include patients who had incident cancer diagnosed from the SEER-Medicare linked database
Sampling Method: Probability Sample
Enrollment: 1132 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-03-29 (Actual)

PRIMARY OUTCOMES:
Incidence of cancer among RA patients treated with abatacept | Approximately 8 years
Incidence of cancer among RA patients treated with anti-TNF's | Approximately 8 years
Incidence of cancer among RA patients treated with other biologics | Approximately 8 years

SECONDARY OUTCOMES:
Incidence of cancer relative to the use of TNFi's in patients taking abatacept | Approximately 8 years
Incidence of cancer relative to the use of other biologic disease modifiers in patients taking abatacept | Approximately 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Princeton, New Jersey, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html